CLINICAL TRIAL: NCT04352101
Title: Effects of Bupropion Versus Escitalopram on Reward Circuitry and Motivational Deficits in Patients With Major Depression and Increased Inflammation and Anhedonia
Brief Title: Bupropion Versus Escitalopram on Reward Circuitry and Motivational Deficits
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Andrew H Miller, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00117673; 1R21MH121891 (NIH)
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Major Depression
Keywords: Inflammation
MeSH Terms: conditions — Depressive Disorder, Major; Inflammation | interventions — Bupropion; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bupropion (Experimental): Participants randomized to take bupropion for 8 weeks.
  Interventions: Drug: Bupropion XL
- Escitalopram (Active Comparator): Participants randomized to take escitalopram for 8 weeks.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Bupropion XL — Participants will take 150 milligrams per day (mg/d) of bupropion XL for two weeks, then the dose will be increased to 300mg/d, as tolerated, for the remaining 6 weeks of the study.
  Other Names: Wellbutrin
  Arms: Bupropion
Drug: Escitalopram — Participants will take 10mg/d of escitalopram for two weeks, then the dose will be increased to 20mg/d, as tolerated, for the remaining 6 weeks of the study.
  Other Names: Lexapro
  Arms: Escitalopram

SUMMARY:
This study is designed to determine whether bupropion (vs escitalopram) increases functional connectivity (FC) within reward-related neurocircuits and decreases motivational deficits in depressed patients with increased inflammation and anhedonia. Participants will be randomized to take bupropion extended release (XL) or escitalopram for 8 weeks.

DETAILED DESCRIPTION:
The goal of the proposed research is to determine the mechanism of action of an antidepressant of known efficacy (bupropion) and to tie this mechanism of action to a biomarker of inflammation in support of precision medicine for the treatment of major depression (MD). MD is a devastating disease affecting approximately 10% of US adults and being the leading cause of disability worldwide. Despite availability of several classes of antidepressant medications, initial treatment response is low (around 30%), and approximately 1/3 of depressed patients are non-responsive to conventional antidepressant therapies. Although extensive reviews of the literature suggest that available antidepressant medications are equally effective, recent studies suggest that there may be differential responsiveness to conventional antidepressants among subgroups of depressed patients. One subgroup of depressed patients who may exhibit differential antidepressant responsiveness are those with increased markers of inflammation. Data from previous studies support the notion that differential responsiveness to conventional antidepressants exists and may be revealed by pretreatment levels of inflammation as indexed by the inflammatory biomarker C-reactive protein (CRP).

This study proposes to use a mechanistic clinical trial design with drugs of known efficacy to take the first step toward establishing whether antidepressants that target dopamine (e.g. bupropion) might be a better choice for depressed patients with increased inflammation and anhedonia than an selective serotonin reuptake inhibitor (SSRI). Accordingly, 50 depressed patients with a CRP>2mg/L and increased anhedonia will be randomized to 8 weeks of bupropion or escitalopram in order to analyze data from 40 patients (accounting for drop outs). All depressed patients will undergo functional magnetic resonance imaging (fMRI) to examine functional connectivity in reward-related circuits at baseline and 4 and 8 weeks along with objective and clinical assessments of Research Domain Criteria (RDoC) positive (motivational) valence constructs at baseline and 2, 4, 6 and 8 weeks.

The researchers hypothesize that patients who receive bupropion versus escitalopram will exhibit increased functional connectivity between ventral striatum and ventromedial prefrontal cortex in association with decreased motivational deficits and anhedonia.

ELIGIBILITY:
Inclusion Criteria:

* willing and able to give written informed consent
* a primary diagnosis of Diagnostic and Statistical Manual of Mental Disorders (DSM-V) MD, current as diagnosed by the Structured Clinical Interview for DSM-V Axis I Disorders (SCID-V)
* score of ≥16 on the 16-item Quick Inventory of Depressive Symptomatology Self-Report (QIDS-SR)
* off all antidepressant or other psychotropic therapy (e.g. mood stabilizers, antipsychotics, and sedative hypnotics) for at least 4 weeks prior to baseline visit (8 weeks for fluoxetine); concomitant administration of up to 2 mg of clonazepam or its equivalent per day will be allowed, but not within 12 hours of study assessments
* CRP>2mg/L
* Inventory of Depressive Symptomatology (IDS-SR) anhedonia subscale score ≥5

Exclusion Criteria:

* history of any autoimmune disorder
* history of hepatitis B or C infection or human immunodeficiency virus infection
* history of any type of cancer requiring treatment with more than minor surgery
* unstable cardiovascular, endocrinologic, hematologic, hepatic, renal, or neurologic disease (as determined by physical examination and laboratory testing)
* history of any (non-mood-related) psychotic disorder; active psychotic symptoms of any type; substance abuse/dependence within 6 months of study entry (as determined by SCID)
* an active eating disorder or antisocial personality disorder
* a history of a cognitive disorder or ≤28 on the Mini-Mental State Exam unless otherwise approved by the PI
* pregnancy or lactation
* chronic use of non-steroidal anti-inflammatory agents (NSAIDS) (excluding 81mg of aspirin), glucocorticoid containing medications
* use of NSAIDS or oral glucocorticoids at any time during the study
* any contraindication for MRI scanning
* failure of more than 2 antidepressant trials in the current episode
* Intolerance of bupropion or escitalopram
* BMI >40 (to exclude severe obesity)
* due to the high co-morbidity between anxiety disorders and depression, the study team plans to include patients with anxiety-related disorders excluding obsessive-compulsive disorder (OCD) if depression is the primary diagnosis. Patients with stable medical conditions and on medications for those conditions will not be excluded. Concomitant administration of up to 2 mg of clonazepam or its equivalent per day will be allowed, but not within 12 hours of study assessments.
* sexually active participants are required to use medically approved birth control methods as defined in the Birth Control Method Form for the duration of the study

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Miller, MD, Principal Investigator — Emory University
Locations (1):
- Emory Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The database generated by the study will be made available to the broader research community upon request accompanied by documentation of local institutional review board (IRB) approval. Investigators will provide relevant protocols and published phenotypic and clinical data upon request.
Supporting Information: Study Protocol
Time Frame: Data will become available two years after the publication of the main findings from the study.
Access Criteria: Material transfers will be made with no more restrictive terms than in the Simple Letter Agreement (SLA) or the Uniform Biological Materials Transfer Agreement (UBMTA) and without reach through requirements. Should any intellectual property arise which requires a patent, the researchers will ensure that the technology (materials and data) remains widely available to the research community in accordance with University policies and the NIH Principles and Guidelines document. A variety of models for data sharing may be adopted, including both central databases and peer-to-peer solutions. Appropriate de-identification techniques should allow sharing of human data, while maintaining appropriate privacy required by both HIPAA and the Common Rule. In addition, informed consent documents should provide sufficient detail about the intent to archive, share and re-analyze data (and samples). Decisions about sharing materials will be made by the study PIs.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Emory Clinic in Atlanta, Georgia, USA. Participant enrollment began September 23, 2020 and the final follow-up assessment occurred July 25, 2022.
Groups:
- Bupropion: Participants randomized to take bupropion for 8 weeks. Participants took 150 milligrams per day (mg/d) of bupropion extended release (XL) for two weeks, then the dose increased to 300mg/d, as tolerated, for the remaining 6 weeks of the study.
- Escitalopram: Participants randomized to take escitalopram for 8 weeks. Participants took 10mg/d of escitalopram for two weeks, then the dose increased to 20mg/d, as tolerated, for the remaining 6 weeks of the study.
Period: Overall Study
Arm/Group | Bupropion | Escitalopram
Started | 10 | 8
Completed | 8 | 7
Not Completed | 2 | 1
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Bupropion: Participants randomized to take bupropion for 8 weeks. Participants took 150 milligrams per day (mg/d) of bupropion XL for two weeks, then the dose increased to 300mg/d, as tolerated, for the remaining 6 weeks of the study.
- Total: Total of all reporting groups
Arm/Group | Bupropion | Escitalopram | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (10.0) | 41.5 (10.3) | 40.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 9 | 7 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Targeted Ventromedial Prefrontal Cortex-Ventral Striatal (vmPFC-VS) Functional Connectivity (FC)
Description: Targeted FC is calculated as the degree of correlation in activity between a 3mm3 radius sphere in VS and the vmPFC cluster identified as being reward-sensitive in neuroimaging meta-analyses and as used to define vmPFC in previous work. Subject-level correlations for degree of vmPFC-VS FC is Fisher's Z transformed {Z(R)=0.5ln[(1+R)/(1-R)]}, a standard method for calculating fMRI functional connectivity, whereby greater Z-scores reflected stronger correlated functional magnetic resonance imaging (fMRI) activity (i.e., higher VS-vmPFC connectivity). For each study timepoint, Z-scores will be extracted and the change in mean FC values compared to baseline will be calculated. The central value is 0, and the standard deviation depends on the sample variance. Increasing values indicate increasing connectivity between the indicated brain regions (VS and vmPFC). There are no relevant thresholds, and there is no direct interpretation of results in terms of clinical improvement.
Time Frame: Baseline, Week 4, Week 8
Population: This analysis includes participants with available and analyzable fMRI scans both at baseline and post-treatment.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Bupropion | Escitalopram
Number analyzed (Participants) | 7 | 5
Z-score
  Baseline to Week 4: number analyzed (Participants) | 7 | 4
  Baseline to Week 4 | 0.02 (0.14) | -0.13 (0.16)
  Baseline to Week 8 | 0.02 (0.20) | 0.09 (0.19)

2. Secondary Outcome: Proportion of Hard-Task Choices During the Effort-Expenditure for Rewards Task (EEfRT)
Description: The Effort-Expenditure for Rewards Task (EEfRT) is a computer-based multi-trial game to assess motivation. Participants are given an opportunity to choose different task difficulty levels to obtain monetary rewards (easy tasks have low rewards while hard tasks have higher rewards). Each trial has a high, medium, or low probability of success, and this information is given to the participant when they are deciding between easy and hard tasks. The task lasts for 20 minutes, and first 50 trials are analyzed. The proportion of hard-task choices across each level of probability is calculated. Possible values range between 0 to1 with 1 being a better outcome indicating the mean probability of making a hard (high effort) choice. Lower proportions of hard task choices indicate decreased motivation.
Time Frame: Baseline, Week 2, Week 4, Week 8
Population: One participant in the Bupropion group was excluded prior to completing this task, and another did not complete the task due to shoulder pain during the task. One participant in the Escitalopram group did not complete the task at the Week 4 visit because the visit was seen virtually (due to illness) and neuropsychological testing was not performed.
Measure: Mean (Standard Deviation); unit: proportion of hard-task choices
Arm/Group | Bupropion | Escitalopram
Number analyzed (Participants) | 8 | 8
proportion of hard-task choices
  Baseline | 0.392 (0.257) | 0.450 (0.290)
  Week 2 | 0.450 (0.316) | 0.385 (0.275)
  Week 4: number analyzed (Participants) | 8 | 7
  Week 4 | 0.348 (0.207) | 0.321 (0.215)
  Week 8: number analyzed (Participants) | 8 | 7
  Week 8 | 0.360 (0.229) | 0.323 (0.158)

3. Secondary Outcome: Snaith-Hamilton Pleasure Scale (SHAPS-C) Score
Description: The SHAPS-C is a 14-item clinician-administered scale assessing the amount of pleasure during common daily activities that the participant has experienced in the past week. Responses are given on a scale of 1 to 4 where 1 = lots of pleasure and 4 = no pleasure. Total scores range from 14 to 56 with lower scores indicating greater enjoyment of activities.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: This analysis includes participants who were still participating in the study at the indicated study visit.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Bupropion | Escitalopram
Number analyzed (Participants) | 10 | 8
Score on a scale
  Baseline | 39.400 (6.535) | 38.625 (2.200)
  Week 2: number analyzed (Participants) | 9 | 8
  Week 2 | 36.222 (6.629) | 33.375 (4.534)
  Week 4: number analyzed (Participants) | 9 | 8
  Week 4 | 33.778 (9.680) | 27.250 (3.196)
  Week 6: number analyzed (Participants) | 8 | 8
  Week 6 | 35.375 (7.963) | 25.250 (4.559)
  Week 8: number analyzed (Participants) | 8 | 7
  Week 8 | 32.125 (9.125) | 24.857 (6.890)

4. Secondary Outcome: Motivation and Pleasure Scale-Self-Report (MAP-SR) Score
Description: The MAP-SR is an 18-item self-report inventory that has been validated in psychiatric populations and is designed to disentangle motivational and consummatory components of everyday activities over a 24-hr period. Responses are given on a 5-point scale where 0 = no pleasure or motivation and 4 = extreme pleasure or motivation. Total scores range from 0 to 72 and higher scores indicate greater motivation and pleasure during everyday activities.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: This analysis includes participants who were still participating in the study at the indicated study visit. One participant in the Bupropion group did not complete this assessment at the Week 4 visit.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Bupropion | Escitalopram
Number analyzed (Participants) | 10 | 8
Score on a scale
  Baseline | 27.800 (7.829) | 28.000 (8.211)
  Week 2: number analyzed (Participants) | 9 | 8
  Week 2 | 29.333 (8.846) | 34.875 (8.493)
  Week 4: number analyzed (Participants) | 8 | 8
  Week 4 | 35.250 (9.254) | 42.500 (11.199)
  Week 6: number analyzed (Participants) | 8 | 8
  Week 6 | 37.250 (8.876) | 44.750 (9.852)
  Week 8: number analyzed (Participants) | 8 | 7
  Week 8 | 38.000 (10.529) | 45.714 (9.232)

5. Secondary Outcome: Inventory of Depressive Symptomatology - Self-Report (IDS-SR)
Description: The IDS-SR is a 30-item self-reported measurement of depression severity. Responses are given on a 4-point scale where 0 = no problems and 3 = severe problems. Total scores are based on 28 items and range from 0 to 84 with higher scores indicating more severe symptoms of depression.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: This analysis includes participants who were still participating in the study at the indicated study visit.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Bupropion | Escitalopram
Number analyzed (Participants) | 10 | 8
Score on a scale
  Baseline | 38.800 (9.942) | 42.250 (7.906)
  Week 2: number analyzed (Participants) | 9 | 8
  Week 2 | 30.222 (8.729) | 30.250 (9.407)
  Week 4: number analyzed (Participants) | 9 | 8
  Week 4 | 23.556 (11.577) | 21.500 (9.258)
  Week 6: number analyzed (Participants) | 8 | 8
  Week 6 | 25.000 (11.464) | 16.250 (11.235)
  Week 8: number analyzed (Participants) | 8 | 7
  Week 8 | 23.875 (11.532) | 18.143 (12.734)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the baseline assessment and continued through the final assessment at Week 8.
Arm/Group | Bupropion | Escitalopram
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 6/10 | 6/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bupropion (N=10) | Escitalopram (N=8)
Nocturnal perspiration (Endocrine disorders) | 1 | 0
Itching (Skin and subcutaneous tissue disorders) | 2 | 0
Lightheadedness (General disorders) | 1 | 0
Headache (General disorders) | 1 | 1
Dry mouth (General disorders) | 1 | 0
Chest pain (Cardiac disorders) | 1 | 0
High blood pressure (Vascular disorders) | 1 | 0
Enlarged lymph nodes (Blood and lymphatic system disorders) | 1 | 0
Pain in limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Stress (Psychiatric disorders) | 1 | 0
Insomnia (General disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3
Vivid dreams (General disorders) | 1 | 0
Anxious mood (Psychiatric disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Sleep disturbance (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 2
Drowsiness (General disorders) | 0 | 1
Tightness in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Nightmares (General disorders) | 0 | 1
Decreased libido (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/01/NCT04352101/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/01/NCT04352101/ICF_001.pdf